CLINICAL TRIAL: NCT04831268
Title: Effects of Traditional Greek Meals: Lentils With Lupino, Trahanas With Tomato Sauce and Halva With Currants on Glycemic Responses: Randomized Clinical Trial in Healthy Humans
Brief Title: Effects of Traditional Greek Meals on Glycemic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HRBD 24 04/04/2019
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; lentils; trahanas; halva; glycemic index
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glucose as reference food (Experimental): Twelve healthy, normal weight subjects (male: 7, female:
  7) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from lentils and lupins, trahanas with tomato sauce and halva with currants, tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Lentils and lupins mixed meal; Other: Trahanas with tomato sauce mixed meal; Other: Halva with currants mixed meal
- Lentils and lupins mixed meal (Experimental): Twelve healthy, normal weight subjects (male: 7, female:
  7) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from lentils and lupins, trahanas with tomato sauce and halva with currants, tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Lentils and lupins mixed meal; Other: Trahanas with tomato sauce mixed meal; Other: Halva with currants mixed meal
- Trahanas with tomato sauce mixed meal (Experimental): Twelve healthy, normal weight subjects (male: 7, female:
  7) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from lentils and lupins, trahanas with tomato sauce and halva with currants, tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Lentils and lupins mixed meal; Other: Trahanas with tomato sauce mixed meal; Other: Halva with currants mixed meal
- Halva with currants mixed meal (Experimental): Twelve healthy, normal weight subjects (male: 7, female:
  7) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from lentils and lupins, trahanas with tomato sauce and halva with currants, tested once, in different weeks along with 250ml water. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: Lentils and lupins mixed meal; Other: Trahanas with tomato sauce mixed meal; Other: Halva with currants mixed meal

INTERVENTIONS:
Other: Glucose as reference food — Twelve healthy, normal weight subjects (male: 7, female:7) after 10-14 hr fast, consumed 25g glucose diluted in 250ml water, tested three times, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were takenat baseline, 15, 30, 45, 60, 90 and 120min.
Other: Lentils and lupins mixed meal — Twelve healthy, normal weight subjects (male: 7, female:7) after 10-14 hr fast, consumed 25g available carbohydrates from lentils and lupins mixed meal along with 250ml water, tested once, in different weeks, within 10-15min. Fingertip capillary blood glucose samples were takenat baseline, 15, 30, 45, 60, 90 and 120min.
Other: Trahanas with tomato sauce mixed meal — Twelve healthy, normal weight subjects (male: 7, female:7) after 10-14 hr fast, consumed 25g available carbohydrates from trahanas with tomato sauce mixed meal along with 250ml water, tested once, in different weeks, within 10-15min. Fingertip capillary blood glucose samples were takenat baseline, 15, 30, 45, 60, 90 and 120min.
Other: Halva with currants mixed meal — Twelve healthy, normal weight subjects (male: 7, female:7) after 10-14 hr fast, consumed 25g available carbohydrates from halva with currants mixed meal along with 250ml water, tested once, in different weeks, within 10-15min. Fingertip capillary blood glucose samples were takenat baseline, 15, 30, 45, 60, 90 and 120min.

SUMMARY:
This study investigated the effects of Greek traditional meals in dehydrated form consumed after reconstitution with water on glycemic responses

DETAILED DESCRIPTION:
This study aimed at 1. to determined the glycemic index and glycemic load of three mixed meals and 2. to investigate the effects of these mixed meals on postprandial glycemic response in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* non-diabetic men and women
* normal body mass index (BMI; between 18.5 and 25 kg/m2)

Exclusion Criteria:

* severe chronic disease (e.g. coronary heart disease, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol
* drug dependency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120 min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g hunger, satiety, desire to eat etc.
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2hr after consumption of three mixed meals

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece